CLINICAL TRIAL: NCT06890312
Title: Timing of Anticoagulant Administration During Radial Access Percutaneous Coronary Intervention: the HERA-PCI Study (Heparin Early for Radial Access Percutaneous Coronary Intervention)
Acronym: HERA-PCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 9323
Record Dates: First submitted 2024-07-16; First posted 2025-03-24 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Coronary Angiography; Percutaneous Coronary Intervention; Radial Artery Occlusion; Bleeding; Anticoagulation
Keywords: Anticoagulant injection timing; Percutaneous coronary intervention; Coronary angiography; Radial artery occlusion prevention; Bleeding events
MeSH Terms: conditions — Arterial Occlusive Diseases; Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "heparin delayed injection" (Active Comparator): Administration of heparin after sheath insertion
  Interventions: Procedure: Administration of heparin after sheath insertion
- heparin early injection (Experimental): Administration of heparin prior to sheath insertion
  Interventions: Procedure: Administration of heparin prior to sheath insertion

INTERVENTIONS:
Procedure: Administration of heparin after sheath insertion — Administration of heparin after sheath insertion
  Arms: "heparin delayed injection"
Procedure: Administration of heparin prior to sheath insertion — Administration of heparin prior to sheath insertion
  Arms: heparin early injection

SUMMARY:
While the reduced hemorrhagic risk of radial access for percutaneous coronary intervention compared to femoral access is well-established, its main complication remains radial artery occlusion, which can occur in up to 30% of patients. Anticoagulation is the primary preventive measure recommended in clinical practice to reduce the risk of this complication, typically involving heparin injection during the procedure in most centers. However, data on the effect of the timing of heparin injection are limited. The investigators hypothesize that injection of heparin before sheath insertion may reduce the rate of radial artery occlusion compared with injection after sheath insertion.

DETAILED DESCRIPTION:
Prevention of radial occlusion relies on optimal hemostasis and anticoagulation. Previous studies have demonstrated a decrease incidence of radial artery occlusion through hemostasis at the puncture site using short-duration mechanical compression methods, guided by mean arterial pressure measurement, or clinical tests evaluating hand vascularization. Anticoagulation plays a central role in the prevention of radial occlusion. It is currently recommended to administer a systemic anticoagulant during a procedure using radial access. Despite the lack of consensus on the nature of the anticoagulant, an international survey showed that more than 90% of interventional cardiologists use unfractionated heparin. The intensity of anticoagulation is also associated with the risk of radial artery occlusion, with previous studies showing that the risk is reduced with the use of "high doses" (5000 IU or 75 IU/kg) compared to "low doses" (<5000 IU or <50 IU/kg). A randomized controlled trial did not show any difference between intravenous and intra-arterial heparin injection via the sheath. No studies have examined the timing of anticoagulant administration relative to sheath insertion. In current practice, anticoagulant administration is typically done after sheath insertion in the radial artery. This common practice likely stems from historical concerns about conversion to femoral access (which is now rare due to improved devices for radial puncture and less consequential due to vascular closure systems used in femoral access, significantly reducing hemorrhagic risk).

No data is currently available on the optimal timing of anticoagulant administration, despite the potential modification of its local effect if the sheath is already in place in the radial artery during the anticoagulant injection, obstructing the radial artery lumen. Our hypothesis is that intravenous anticoagulant administration before sheath insertion in the radial artery is more effective than administration after sheath insertion in patients undergoing percutaneous coronary intervention via radial access. The expected outcomes include a reduction in the incidence of radial artery occlusion after the procedure, leading to a decrease in potential complications (acute hand ischemia, failure of the access route during a subsequent procedure, inability to create an ipsilateral arteriovenous fistula).

The primary objective is to evaluate the impact of the timing (early or late) of intravenous anticoagulant administration on the risk of radial occlusion during a percutaneous coronary intervention via radial access.

This is a single-center, comparative, randomized, single-blind study with blinded evaluation of the primary endpoint.

After providing information and verifying eligibility criteria, the investigator will obtain the patient's free, informed, and written consent before any intervention, on the day the coronary angiography is scheduled. Consent will be obtained in the patient's hospital room (Cardiology Day Hospital or conventional hospitalization unit).

Randomization, in blocks of variable sizes, will be carried out by the investigator (or a delegate) after consent is signed and eligibility criteria are verified and before the percutaneous coronary intervention via radial access. Randomization assigns the subject's inclusion number and treatment group:

* Control group "delayed injection": administration of heparin after sheath insertion
* Experimental group "early injection": administration of heparin before sheath insertion Randomization will be done via a centralized electronic system called Cleanweb.

The percutaneous coronary intervention via radial access will be performed according to standard practice in the cardiac catheterization lab of our center. At the time of installation, the operator will palpate the radial pulse to ensure the feasibility of radial access. In the experimental group "early injection" of heparin, the injection will be done intravenously just before skin disinfection, approximately 5 minutes (± 3 minutes) before the puncture. In the control group "delayed injection", the injection will be done 5 minutes (± 3 minutes) after sheath insertion into the radial artery (protocol used in daily practice). If radial puncture fails, patients will be excluded from the primary endpoint analysis but will be followed up at 30 days for secondary endpoints. The heparin bolus dose will systematically be 50 IU/kg. At the end of the procedure, an ACT will be measured just before sheath removal, and hemostasis at the puncture site will be achieved using a TR-band® mechanical compression device. This will be placed before sheath removal and inflated with a syringe containing 15 cc of air for all patients. According to local protocol, mechanical compression is left in place for 2 hours before gradual deflation (removal of 2 cc every 15 minutes until complete deflation, bracelet left in place for 30 minutes post-deflation, then removed and replaced with a simple dressing). In case of additional coronary angioplasty, the heparin dose will be adjusted based on the angioplasty indication at the operators' discretion for a total dose of 0.7 to 1.0 mg/kg, aiming for an ACT > 250 ms.

At day 1, the following will be performed according to standard practice:

* An interview
* A clinical examination
* An upper limb arterial Doppler ultrasound on the same side as the radial puncture

At day 30 (±7 days), patients will be contacted by phone specifically for the research by the investigators and co-investigators involved in the study. The telephone interview will consist of an inquiry for symptoms of radial occlusion or major cardiovascular events. If symptoms of radial occlusion are detected, the patient will be scheduled for a consultation with a clinical examination, pulse palpation, Barbeau maneuver, and upper limb arterial Doppler ultrasound on the same side as the radial puncture.

The primary endpoint is the rate of radial artery occlusion, as determined by Doppler ultrasound at day 1.

The secondary endpoints are:

* The rate of symptomatic radial artery occlusion (acute hand ischemia) on day 1. The rate of occlusion will be assessed through a thorough clinical examination on day 1 after the procedure, and if necessary, based on clinical findings, by an upper limb CT angiography. A telephone interview will also be conducted on day 30 to check for symptoms of symptomatic radial artery occlusion (signs of hand ischemia). If symptoms are present, the patient will be scheduled for a consultation with arterial Doppler ultrasound to confirm or rule out radial occlusion.
* Major cardiovascular events within the first 30 days following the percutaneous coronary intervention: cardiovascular death, myocardial infarction, and stroke. These events will be assessed during the visits on day 1 and day 30.
* Local hemorrhagic events assessed by checking for a hematoma of at least 2 cm on day 1 and general hemorrhagic events evaluated on day 30 according to the BARC (Bleeding Academic Research Consortium) classification.
* Local functional impact evaluated on day 30 by the presence of residual pain in the radial region or limited joint mobility.
* The rate of radial puncture failure.
* The occurrence of all-cause mortality on day 30.

ELIGIBILITY:
Inclusion Criteria:

* Patients having 18 years old or older, regardless of gender, undergoing percutaneous radial coronary intervention
* Subject affiliated to a social protection health insurance
* Subject able to understand the objectives and risks of the research and to provide dated and signed consent
* Subject who has been informed of the results of the preliminary medical examination

Exclusion Criteria:

* Contraindication to the use of heparin (history of heparin-induced thrombocytopenia)
* Very high bleeding risk defined by recent bleeding (<6 months) of type 3 of the BARC classification
* Subject in an exclusion period (determined by a previous or ongoing study)
* Inability to give the subject enlightened information (subject in an emergency situation, difficulties in understanding the subject, etc.)
* Subject under safeguard of justice
* Subject under guardianship or curatorship
* Pregnancy
* Breastfeeding
* Patient on anticoagulant treatment: anti-vitamin K, direct oral anticoagulants (DOACs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Rate of radial artery occlusion | Day 1
  The primary endpoint is the rate of radial artery occlusion, as determined by Doppler ultrasound at day 1.

SECONDARY OUTCOMES:
Rate of symptomatic radial artery occlusion (acute hand ischemia) on day 1 | Day1
  The rate of symptomatic radial artery occlusion (acute hand ischemia) on day 1. The rate of occlusion will be assessed through a thorough clinical examination on day 1 after the procedure, and if necessary, based on clinical findings, by an upper limb CT angiography. A telephone interview will also be conducted on day 30 to check for symptoms of symptomatic radial artery occlusion (signs of hand ischemia). If symptoms are present, the patient will be scheduled for a consultation with arterial Doppler ultrasound to confirm or rule out radial occlusion.
Major cardiovascular events within the first 30 days following the percutaneous coronary intervention: cardiovascular death, myocardial infarction, and stroke. | Day 30
  Major cardiovascular events within the first 30 days following the percutaneous coronary intervention: cardiovascular death, myocardial infarction, and stroke. These events will be assessed during the visits on day 1 and day 30
Local and general hemorrhagic events | Day 30
  Local functional impact evaluated on day 30 by the presence of residual pain in the radial region or limited joint mobility.
Rate of radial puncture failure. | Day 0
  The rate of radial puncture failure.
Rate of all-cause mortality on day 30. | Day 30
  The occurrence of all-cause mortality on day 30.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, Bas-Rhin, France

IPD SHARING:
Plan to Share IPD: No